CLINICAL TRIAL: NCT02079857
Title: Symptom Management for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-02325; R01NR013695 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Standard (Experimental): Fixed protocol
  Interventions: Other: Standard protocol
- Individualized (Experimental): Individualized protocol
  Interventions: Other: Individualized protocol
- Control (Sham Comparator): Sham acupuncture/Placebo moxa
  Interventions: Other: Sham acupuncture/Placebo moxa

INTERVENTIONS:
Other: Standard protocol — Subjects will receive a standard treatment
  Arms: Standard
Other: Individualized protocol — Subjects will receive an individualized treatment
  Arms: Individualized
Other: Sham acupuncture/Placebo moxa — Subjects will receive sham acupuncture/placebo moxa
  Arms: Control

SUMMARY:
The objective of this study is to test the efficacy of a symptom management treatment strategy, Acupuncture/Moxibustion (Acu/Moxa), to improve the symptoms associated with Irritable Bowel Syndrome (IBS) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 70 years of age.
* Diagnosis of IBS based on ROME III criteria.
* Complete symptom diaries and return completed diaries at all sessions.

Exclusion Criteria:

* History of co-existing gastrointestinal, and/or gynecological, and/or urologic pathology.
* Alarm symptoms according to ROME III.
* Individuals currently receiving other types of complementary therapies.
* Individuals with an acute medical condition requiring acute medical attention.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Symptom severity-abdominal pain | week 1
Symptom severity-abdominal pain | week 4
Symptom severity-abdominal pain | week 8
Symptom severity-abdominal pain | week 12
Symptom severity-abdominal pain | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Anastasi, PhD, Principal Investigator — New York University
Locations (1):
- NYU Division of Special Studies in Symptom Management, New York, New York, United States